CLINICAL TRIAL: NCT04683484
Title: Clinical Trials of Phase 1, 2 of Nanocovax Manufactured by Nanogen
Brief Title: A Clinical Trial to Assess the Safety and Immunogenicity of Nanocovax in Heathy Volunteers
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanogen Pharmaceutical Biotechnology Joint Stock Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NNG26
Record Dates: First submitted 2020-12-18; First posted 2020-12-24 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low dose of Nanocovax (Experimental): Intramuscular injection, two doses given 28 days apart
  Interventions: Biological: Nanocovax
- Middle dose of Nanocovax (Experimental): Intramuscular injection, two doses given 28 days apart
  Interventions: Biological: Nanocovax
- High dose of Nanocovax (Experimental): Intramuscular injection, two doses given 28 days apart
  Interventions: Biological: Nanocovax
- Placebo (Placebo Comparator): Intramuscular injection, two doses given 28 days apart
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Nanocovax — Recombinant Protein spike (s) SARS-CoV-2 and adjuvant (0,5 mg Al PO4)
  Arms: High dose of Nanocovax; Low dose of Nanocovax; Middle dose of Nanocovax
Biological: Placebo — 0,5 mg Al PO4
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety, tolerability, and immunization of Nanocovax in healthy volunteers.

DETAILED DESCRIPTION:
The clinical trial Phase 1, open-label, dose-escalation to evaluate the safety, tolerability, and initial assessment of immunogenicity of the vaccine Nanocovax intramuscularly in healthy Vietnamese adult volunteers.

The clinical trial Phase 2, randomization, double-blind, multicenter, placebo-controlled to evaluate the safety, immunogenicity, and determined the optimal dose of the Vaccine Nanocovax intramuscularly in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* From 18 to 50 years old in phase 1, from 12 to 75 years old in phase 2
* Body Mass Index (BMI) between 18 and 28 kg/m2
* The subject has good health, is assessed through medical history, clinical examination, and laboratory tests (such as hematology, biochemistry, urine ...) within the normal range evaluated by the clinician.
* Subjects aged potentially pregnant should use effective contraceptive methods 4 weeks prior to screening and during the study and last until 6 months after the last injection.
* Able and willing to participate in all activities in the clinical trial, including 6-month follow-up after vaccination.
* Sign the consent form. For a subject from 12 to 17 years old, it is necessary to have a legal guardian sign the consent form to participate in the study

Exclusion Criteria:

* Insufficient civil act capacity.
* Subjects at high risk of SARS-CoV-2 infection.
* Subject is/has ever had any acute or chronic medical condition, including but not limited to:

  * Have any inflammatory disease, respiratory tract infection, have any respiratory symptoms such as: cough, sore throat, difficulty breathing, wheezing due to respiratory symptoms within 07 days before screening. Fever (armpit temperature ≥ 37°C) for 3 days before vaccination.
  * History of any chronic respiratory illness such as bronchial asthma, chronic bronchitis, cystic fibrosis, chronic obstructive pulmonary disease (COPD).
  * Malignant disease
  * Immune disorders, using immunosuppressive therapy.
  * Cardiovascular diseases (including high blood pressure requiring drug treatment), liver disease, chronic kidney disease, endocrine diseases (including diabetes), hemoglobin disease ...
  * Neurological, psychiatric, epilepsy, or Guillian-Barré disorders.
  * Pathology of hemostasis.
  * Having any surgery for 8 weeks before screening.
  * History of organ transplantation.
* Examination and testing results at the time of screening:

  * Systolic pressure above 140 mmHg and/or diastolic pressure over 90mmHg;
  * Systolic blood pressure less than 90 mmHg and/or diastolic pressure below 50 mmHg
  * Real-Time nasopharyngeal fluid test - PCR (positive) and/or anti S - IgG (positive) with SARS-CoV-2.
  * Women of potential pregnancy, a positive urine beta-hCG test at the time of screening.
  * Positive with HIV, hepatitis B (HBsAg), hepatitis C (ANTI-HCV) tests
  * WBC less than 3.5 x 10^9 cells / L
  * Lymphocytes of less than 1.0 x 10^9 cells / L.
  * Neutrophils less than 2.0 x 10^9 cells / L
  * Platelets below 140 x 10^9 cells / l
  * Hb less than 120 g/L for men and less than 100 g/L for women
  * ALT or AST is over 2 times the normal limit
  * eGFR of 90 mL/min/ 1.73m2 or less.
  * Abnormal ECG of clinical significance.
* The Subject who have taken any drugs or treatments simultaneously and before:

  * Any drug or treatment that affects the immune system such as injectable anti-allergenic drugs, Globulin, Interferon, immunomodulators, cytotoxic drugs, or any other drug toxic to the body, for 90 days before screening.
  * Systemic steroids (oral or injectable; including intra-articular injection) regardless of dose except for topical form, for 28 days prior to screening.
  * Any vaccine within 28 days prior to screening or planned for in-study vaccination or after 6 months after the first vaccination.
  * Receive or donate blood/serum during the 8 weeks prior to the screening, or plan to receive or donate blood/serum during the study period.
* The Subject that participated in any clinical trial 28 days prior to the screening date or intends to participate in another clinical study at any point in the study.
* Women who are pregnant and breastfeeding or planning to become pregnant for the next 6 months from the time of the study 2 vaccines.
* The Subject has a history of allergy to any of the vaccine components understudying or has a history of at least one past history of allergic or hypersensitivity reactions.
* The Subject addicted to alcohol (drinking from 5 cups of alcohol daily, glasses of alcohol/can of beer), tobacco/water pipe addicts (smoking from 5 or more cigarettes), drug addiction, opioid dependence
* The Subject is a member of the research team, sponsor employee, producer (Nanogen), and a person related by family (wife, husband, child, father, mother) with those subjects.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 620 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-06-10 (Estimated); Study Completion 2021-08-10 (Estimated)

PRIMARY OUTCOMES:
Solicited adverse events | 7 days after each dose
  Percentage and severity level of participants reporting Solicited adverse events
Anti-S IgG | 0, 7, 28, 35, 56, 180 days after the first dose
  Geometric mean concentrations of Anti-S IgG at each time points

SECONDARY OUTCOMES:
SARS-CoV-2 neutralizing titers | 0, 7, 28, 35, 56, 180 days after the first dose
  Geometric mean titers of SARS-CoV-2 Neutralization antibody at each time points
Participants achieving ≥4-fold rise of Anti-S IgG | 0, 7, 28, 35, 56, 180 days after the first dose
  Proportion of participants achieving ≥4-fold rise of Anti-S IgG from before vaccination at each time points
Cellular immune response (IFNγ) | 28, 35, 56 days after the first dose
  Change of IFNγ from baseline after vaccination
Cellular immune response (T CD4) | 28, 35, 56 days after the first dose
  Change of T CD4 from baseline after vaccination
Cellular immune response (T CD8) | 28, 35, 56 days after the first dose
  Change of T CD8 from baseline after vaccination
Serious adverse events | 28 days after each dose
  Percentage of participants reporting Serious adverse events
Unsolicited adverse events | 28 days after each dose
  Percentage of participants reporting Unsolicited adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Military Medical Academy, Hanoi, Ha Dong, Vietnam

REFERENCES:
- [Derived] Nguyen TP, Do Q, Phan LT, Dinh DV, Khong H, Hoang LV, Nguyen TV, Pham HN, Chu MV, Nguyen TT, Pham QD, Le TM, Trang TNT, Dinh TT, Vo TV, Vu TT, Nguyen QBP, Phan VT, Nguyen LV, Nguyen GT, Tran PM, Nghiem TD, Tran TV, Nguyen TG, Tran TQ, Nguyen LT, Do AT, Nguyen DD, Ho SA, Nguyen VT, Pham DT, Tran HB, Vu ST, Hoang SX, Do TM, Nguyen XT, Le GQ, Tran T, Cao TM, Dao HM, Nguyen TTT, Doan UY, Le VTT, Tran LP, Nguyen NM, Nguyen NT, Pham HTT, Nguyen QH, Nguyen HT, Nguyen HLK, Tran VT, Tran MTN, Nguyen TTT, Ha PT, Huynh HT, Nguyen KD, Thuan UT, Doan CC, Do SM. Safety and immunogenicity of Nanocovax, a SARS-CoV-2 recombinant spike protein vaccine: Interim results of a double-blind, randomised controlled phase 1 and 2 trial. Lancet Reg Health West Pac. 2022 May 16;24:100474. doi: 10.1016/j.lanwpc.2022.100474. eCollection 2022 Jul. PMID 35602004